CLINICAL TRIAL: NCT04562714
Title: IMpact of Flash Glucose Monitoring in pEople With Type 2 Diabetes Inadequately Controlled With Non-insulin Antihyperglycemic ThErapy - IMMEDIATE Study
Brief Title: Impact of Flash Glucose Monitoring in People With Type 2 Diabetes Using Non-Insulin Antihyperglycemic Therapy
Acronym: IMMEDIATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IMMEDIATE
Record Dates: First submitted 2020-09-01; First posted 2020-09-24 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2; Glucose
Keywords: Type 2 diabetes; Flash sensor glucose technology; Glucose monitoring; Randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The IMMEDIATE study is a two-phased, cross-over study. In Phase 1, participants will be randomized at a 1:1 ratio, stratified by use of glucagon-like peptide-1 receptor agonist to receive either a flash glucose monitor (FGM) + diabetes self-management education (DSME) (Intervention arm) or to DSME alone (Control arm). Participants randomized to the Intervention arm will receive a FreeStyle Libre FGM System, 1 training session on its proper use, and 6 DSME sessions. Participants randomized to the Control arm will receive 6 DSME sessions matched to time and location of the Intervention group. DSME sessions for both groups will consist of four individual in-clinic sessions and two telephone sessions. After 16-weeks, participants initially assigned to DSME alone will cross-over to receive the intervention FGM device, while those initially randomized to using a FGM will continue using their device for an additional 16 weeks (Phase 2). No DSME will provided during Phase 2.
Masking Description: The study design is open-label in which neither investigator nor study participants will be blinded to study treatment. All study participants will wear a blinded continuous glucose monitoring device for two weeks at baseline and during the final two weeks of Phase 1, during which they will be blinded to the results of the blinded glucose monitoring device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (FGM + DSME) (Experimental): Study participants randomized to the intervention arm will be provided with a FreeStyle Libre flash glucose monitor (FGM) system to use for 16 weeks in Phase 1. Study participants will receive one training session on proper use of the FGM and encouraged to test at least 4 times per day: fasting and post-meals. Participants will also receive six diabetes self-management education (DSME) sessions, consisting of four individual in-clinic sessions and two telephone sessions.
  Interventions: Device: FreeStyle Libre Flash Glucose Monitor; Other: Diabetes self-management education
- Control (DSME alone) (Other): Study participants in the control arm will receive six diabetes self-management education sessions matched to time and location of the intervention group. The sessions will consist of four individual in-clinic sessions and two telephone sessions over 16 weeks. Control participants will be encouraged to self-monitor blood glucose four times daily (fasting and post-meals) as per existing diabetes self-care guidelines
  Interventions: Other: Diabetes self-management education

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitor — The FreeStyle Libre FGM device consists of a skin-worn disposable sensor that automatically measures and continuously stores glucose readings. The sensor is placed by a single-use applicator and is activated by a wireless scan with a handheld reader. It is designed to stay on the body for up to 14 days, and can be worn under clothing. After a 1-hour warm-up period, the sensor takes automatic measurements of glucose every 15 minutes for up to 14 days. The device collects the interstitial glucose values and stores them for subsequent upload at the end of the 14-day wear period. With each scan, users receive their glucose reading; the last eight hours of glucose data; and an arrow illustrating the direction their glucose is heading.
  Arms: Intervention (FGM + DSME)
Other: Diabetes self-management education — The DSME curriculum is compromised of:
  1. Review of weekly glucose report (Trend glucose report from Libreview for intervention group; and weekly glucose report in log book format from their glucose monitoring software for control group)
  2. Education modules for both in-person and remote delivery;
  3. Handouts to support the curriculum objectives; and
  4. Blood glucose monitoring challenges to stimulate behaviour change and reinforce learning.

SUMMARY:
The objective of this study is to evaluate the effectiveness of a flash glucose monitor device in achieving optimal glycemic control among adults with type 2 diabetes inadequately controlled with non-insulin antihyperglycemic therapy.

DETAILED DESCRIPTION:
The IMMEDIATE study is a multi-centre, randomized controlled, open-label, two-phase cross-over study evaluating the effectiveness of a flash glucose monitor device to increase the proportion of time spent in target glucose range (3.9 to 10.0 mmol/L) among adults with type 2 diabetes inadequately controlled with non-insulin antihyperglycemic therapy compared to a control group not using a flash glucose monitor device. The study will consist of two phases; each 16 weeks long. In Phase 1, study participants who meet eligibility criteria will be randomized to receive a flash glucose monitor device combined with diabetes self-management education, or diabetes self-management education alone. In Phase 2, participants initially assigned to receive education alone will crossover to receive a flash glucose monitor device while participants initially using the flash glucose monitor will continue using their device. No diabetes self-management education will be provided during Phase 2.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must be an adult aged 18 years or older and:

* A clinical diagnosis of T2D, with diagnosis known for six months or more;
* An HbA1c of > 7.5%;
* Using one or more non-insulin antihyperglycemic therapy for a minimum of six months, with dose stability of 3 months; and
* No previous history of using CGM or FGM devices.

Exclusion Criteria:

Participants will be excluded from the study if they:

* Have a history of insulin use > 3 months
* Are pregnant or breastfeeding
* Have diabetic retinopathy
* Have an estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2
* Have unstable cardiovascular disease
* Use other implanted medical devices, such as pacemakers
* Have had more than one episode of severe hypoglycemia during the past 6 months or evidence of hypoglycemia unawareness
* Anticipate or require regular magnetic resonance imaging, computed tomography scan, or high-frequency electrical heat (diathermy) treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Time in Range (TIR) | 2-week period
  The proportion of time within target glucose range (3.9 to 10.0 mmol/L) among adults with type 2 diabetes (T2D) inadequately controlled with non-insulin antihyperglycemic therapy compared to a control group not using an FGM device measured during the blinded continuous glucose monitor (CGM) period during the final last two-weeks of the Phase 1

SECONDARY OUTCOMES:
Glycemic control (a) | 2-week period
  Mean HbA1c (blood drawn for laboratory testing) at the end of Phase 1
Glycemic control (b) | 2-week period
  Proportion of participants with HbA1c < 7.0% and with HbA1c > 9.0% at the end of Phase 1
Glycemic control (c) | 2-week period
  Mean glucose based on blinded CGM recordings at the end of Phase 1
Proportion of time spent in various glycemic ranges based on blinded CGM recordings | 2-week period
  * Tight glycemic range (3.9 to 7.8 mmol/L)
  * Hypoglycemia range (3.0 to 3.8 mmol/L)
  * Clinically significant (level 2) hypoglycemia range (< 3.0 mmol/L)
  * Hyperglycemia (> 10.0 mmol/L)
Glycemic variability | 2-week period
  Standard deviation and % coefficient of variation based on blinded CGM recordings
Number of documented episodes of hypoglycemia episodes | 2-week period
  Based on the blinded CGM recording, including:
  * All (hypoglycemic episode occurring at anytime);
  * Nocturnal (hypoglycemic episode occurring between 12 am and 6 am); and
  * Level 2 hypoglycemic (<3.9 mmol/L)
Number of episodes of severe hypoglycemia | 16-week period
  A hypoglycemic episode that requires assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions as reported by participant
Adherence to diabetes medications as measured by the Adherence to Refills and Medication-Diabetes (ARMS-D) | 2-week period
  The ARMS-D is an 11-item self-reported measure of adherence that assesses one's ability to take and refill medication under different circumstances, and identifies barriers to medication adherence. The ARMS-D demonstrates good internal consistency, reliability (α=0.86), shows good convergent validity with other adherence to medication scales, and independently predicts HbA1c (β=0.16, p<0.01)
Psychological distress as measured by the Diabetes Distress Scale (DDS) | 2-week period
  The DDS is a 17-item scale that captures four dimensions of distress: emotional burden, regime distress, interpersonal distress and physician distress. The DDS list potential problem areas that people with diabetes may experience. Respondents are asked to indicate the degree to which each problem may be bothering them in their life on a 6-point Likert Scale from 1 (not a problem) to 6 (a very serious problem). The DDS and its subscales has been shown to have good internal reliability (α > 0.87) and validity.
Device satisfaction as measured by the Glucose Monitoring System Satisfaction Survey (GMSS) | 2-week period
  The GMSS is a 15-item self-reported measure of glucose device satisfaction. The GMSS provides a comprehensive profile of key contributors to device satisfaction. The GMSS has shown good criterion validity against the World Health Organization-5 measure of quality of life and the DDS, and the Self-Monitoring Blood Glucose (SMBG) Obstacles scale (all p < 0.001)
Participant self-efficacy as measured by the Skills, Confidence and Preparedness Index (SCPI) | 2-week period
  The SCPI is a 23-item scale that includes three subscales: Skills; confidence; and preparedness. Each question contains a 7-point Likert scale response. The SCPI has been demonstrated to have high validity internal consistency and test-retest reliability, with no floor or ceiling effect. Furthermore, SCPI scores are significantly correlated with HbA1c in both type 1 diabetes and T2D populations (p < 0.001)
Change in antihyperglycemic therapies | 2-week period
  Change in the mean number of antihyperglycemic therapies from baseline to end of
Change in weight (kg) | 16-week period
  Change in weight (kg) from baseline to end of Phase 1
Change in waist circumference (cm) | 16-week period
  Change in waist circumference (cm) from baseline to end of Phase 1
Diabetes self-management education (DSME) goals setting | 16-week period
  Mean number of diabetes self-management education (DSME) goals set per person
Mean DSME goal achievement score during Phase 1 | 16-week period
  Each DSME goal set during the trial is be graded on a 6-point rating scale. Goal attainment scores range from 1 (goal not attempted) to 6 (exceeded expectation).
Mean number of glucose checks | 2-week period
  Mean number of FGM scans for the intervention group; and mean number of self-monitoring of blood glucose for the control arm

OTHER OUTCOMES:
Exploratory analysis 1a: Glucose control - Targeted glucose range | 16-week period
  Within group change in the proportion of time spent in targeted glucose range based on FGM metrics from the first 2-week and final 2-week periods of Phase 2
Exploratory analysis 1b: Glucose control - hypoglycemia | 16-week period
  Within group change in the proportion of time spent in hypoglycemia (<3.8 mmol/L) ranged based on FGM metrics from the first 2-week and the final 2-week periods of Phase 2
Exploratory analysis 1c: Glucose control - hyperglycemia | 16-week period
  Within group change in the proportion of time spent in hyperglycemia (>10 mmol/L) range based on FGM metrics from the first 2-weeks and final 2-week periods of Phase 2
Exploratory analysis 1d: Glucose control - HbA1c | 16-week period
  Within group change in HbA1c based on blood drawn for laboratory testing from the first 2-week and the final 2-week periods of Phase 2
Exploratory analysis 1e: Glucose control - Mean glucose | 16-week period
  Within group change in mean glucose based on FGM metrics from the first 2-week and final 2-week periods of Phase 2
Exploratory analysis 1f: Glucose control - Glycemic variability | 16-week period
  Within group change in standard deviation and % coefficient of variation based on FGM metrics from the first 2-week and final 2-week periods of Phase 2
Exploratory analysis 1g: Glucose control - Hypoglycemia | 16-week period
  Within group change in the frequency of hypoglycemia based on FGM metrics from the first 2-week and final 2-week periods of Phase 2
Exploratory analysis 1h: Glucose control - Severe hypoglycemia | 16-week period
  Within group change in the frequency of severe hypoglycemia, defined as a hypoglycemic episode that required assistance of another person to actively administer carbohydrate, glucagon or other resuscitative actions, based on FGM metrics from the first 2-week and final 2-week periods of Phase 2
Exploratory analysis 2a: Patient reported outcome - Adherence | 16-week period
  Within group change in the Adherence to Refills and Medication-Diabetes (ARMS-D) from the beginning to the end of Phase 2
Exploratory analysis 2b: Patient reported outcome - Psychological distress | 16-week period
  Within group change in the Diabetes Distress Scale from the beginning to the end of Phase 2.
Exploratory analysis 2c: Patient reported outcome - Device satisfaction | 16-week period
  Within group change in the Glucose Monitoring System Satisfaction Survey from the
Exploratory analysis 2d: Patient reported outcome - Participant self-efficacy | 16-week period
  Within group change in the Skills, Confidence and Preparedness Index (SCPI) from the beginning to the end of Phase 2.
Exploratory analysis 3a: Effect of DSME goal achievement | 16-week period
  The effect of DSME goal achievement, independent of glucose monitoring system used, on the change in proportion of time spent in targeted glucose range in the final 2-week CGM period of Phase 1 vs baseline
Exploratory analysis 3b: Effect of DSME goal achievement | 16-week period
  The effect of DSME goal achievement, independent of glucose monitoring system used, on the frequency of FGM-measured hypoglycemia in the final 2-week CGM period of Phase 1 vs baseline
Exploratory analysis 3c: Effect of DSME goal achievement | 16-week period
  The effect of DSME goal achievement, independent of glucose monitoring system used, on the association between the daily frequency of FGM scanning/self-monitored blood glucose and TIR.
Exploratory analysis 4: Frequency of glucose testing | 16-week period
  The optimal frequency of glucose testing for greatest impact on glycemic control (TIR)

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, MD, Principal Investigator — LMC Diabetes
Locations (6):
- Canada (6):
  - LMC Brampton, Brampton, Ontario
  - LMC Etobicoke, Etobicoke, Ontario
  - LMC Oakville, Oakville, Ontario
  - LMC Ottawa, Ottawa, Ontario
  - LMC Midtown, Toronto, Ontario
  - LMC Vaughan/Thornhill, Vaughan, Ontario

REFERENCES:
- [Background] Polonsky WH, Fisher L, Hessler D, Edelman SV. Development of a New Measure for Assessing Glucose Monitoring Device-Related Treatment Satisfaction and Quality of Life. Diabetes Technol Ther. 2015 Sep;17(9):657-63. doi: 10.1089/dia.2014.0417. Epub 2015 Apr 29. PMID 25923812
- [Background] Mayberry LS, Gonzalez JS, Wallston KA, Kripalani S, Osborn CY. The ARMS-D out performs the SDSCA, but both are reliable, valid, and predict glycemic control. Diabetes Res Clin Pract. 2013 Nov;102(2):96-104. doi: 10.1016/j.diabres.2013.09.010. Epub 2013 Sep 26. PMID 24209600
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Aronson R, Li A, Brown RE, Walker A, Lyons A, Orzech N. Optimizing Diabetes Self-management Using the Novel Skills, Confidence, and Preparedness Index (SCPI). Diabetes Care. 2019 Oct;42(10):1873-1878. doi: 10.2337/dc19-0699. Epub 2019 Aug 9. PMID 31399439